CLINICAL TRIAL: NCT00434057
Title: Evaluation of Pigmented Skin Lesions With MelaFind(R) System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MELA Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20061
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2009-11-11 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Melanoma
Keywords: Pigmented Skin Lesions; Dermatology; Skin Cancer; Melanoma; MelaFind
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsied Pigmented Skin Lesions (Other): Pigmented skin lesions for which clinical management was prospectively determined to be biopsy of the lesion in toto
  Interventions: Device: MelaFind(R)

INTERVENTIONS:
Device: MelaFind(R) — Biopsy ratio comparison
  Other Names: MF100; MelaFind Device System; MelaFind Device

SUMMARY:
The purpose of this clinical trial is to demonstrate that MelaFind®, a new instrument that uses machine vision for non-invasive early detection of cutaneous pigmented malignant melanoma, is safe and effective. MelaFind® acquires digital images of the lesion with illumination in different spectral bands, from visible to near infrared, and automatically analyzes these images. Diagnostic accuracy of MelaFind® and that of study dermatologists will be evaluated. The reference standard will be final interpretation of lesions by central dermatohistopathology.

ELIGIBILITY:
Inclusion Criteria:

* The lesion is pigmented (i.e., melanin, keratin, blood)
* Clinical management of the lesion by the examining dermatologist is either biopsy of the lesion in toto, or 3-month follow-up of the lesion
* The diameter of the pigmented area is between 2 and 22 millimeters
* The lesion is accessible to the MelaFind hand-held imaging device
* The patient, or a legally authorized representative, has consented to participate in the study and has signed the Informed Consent Form

Exclusion Criteria:

* The patient has a known allergy to isopropyl alcohol
* The lesion has been previously biopsied, excised, or traumatized
* The skin is not intact (e.g., open sores, ulcers, bleeding)
* The lesion is within 1 cm of the eye
* The lesion is on mucosal surfaces (e.g., lips, genitals)
* The lesion is on palmar hands
* The lesion is on plantar feet
* The lesion is on or under nails
* The lesion is located on or in an area of visible scarring
* The lesion contains foreign matter (e.g., tattoo, splinter, marker)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1383 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Gutkowicz-Krusin, PhD, Study Director — Electro-Optical Sciences, Inc.; Joseph V Gulfo, MD, MBA, Study Director — Electro-Optical Sciences, Inc.; Harold S Rabinovitz, MD, Study Chair — Skin and Cancer Associates; Armand B Cognetta, Jr, MD, Study Chair — Dermatology Associates of Tallahassee
Locations (2):
- United States (2):
  - Skin and Cancer Associates, Plantation, Florida
  - Dermatology Associates of Tallahassee, Tallahassee, Florida

REFERENCES:
- [Derived] Monheit G, Cognetta AB, Ferris L, Rabinovitz H, Gross K, Martini M, Grichnik JM, Mihm M, Prieto VG, Googe P, King R, Toledano A, Kabelev N, Wojton M, Gutkowicz-Krusin D. The performance of MelaFind: a prospective multicenter study. Arch Dermatol. 2011 Feb;147(2):188-94. doi: 10.1001/archdermatol.2010.302. Epub 2010 Oct 18. PMID 20956633
- See also: Sponsor Web Site — http://www.eosciences.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Biopsied Pigmented Skin Lesions: Lesions for which clinical management was prospectively determined to be biopsy of the lesion in toto
Period: Overall Study
Arm/Group | Biopsied Pigmented Skin Lesions
Started | 1383
Completed | 1382 (One patient withdrew from the study after signing the Informed Consent Form)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Biopsied Pigmented Skin Lesions
Number analyzed (Participants) | 1383
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56
  Between 18 and 65 years | 1056
  >=65 years | 271
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 745
  Male | 638
Region of Enrollment [Number; unit: participants]
  United States | 1383

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity
Description: Sensitivity is the fraction of correctly identified cases of melanoma. Specificity is the fraction of correctly identified cases of non-melanoma.
Time Frame: Within 120 days of Data Lock
Population: All participants with eligible and evaluable lesions were used in analysis of primary outcome measures
Measure: Mean (95% Confidence Interval); unit: Ratio * 100
Arm/Group | Biopsied Pigmented Skin Lesions
Number analyzed (Participants) | 1257
Ratio * 100
  MelaFind sensitivity to melanoma | 98.2 [95.1 to 100]
  MelaFind specificity for melanoma | 9.5 [6.1 to 12.9]
Statistical Analysis 1: Comparison: Biopsied Pigmented Skin Lesions; MelaFind's sensitivity to cutaneous melanoma and 95% confidence intervals were determined; Test type: Superiority or Other; p = 0.05, exact mid-P; Sensitivity to melanoma = 98, 95% CI [95.1 to 100] — Of 127 melanomas, 114 melanomas had a pre-biopsy diagnosis of "Melanoma can not be ruled out" or "Not melanoma," which qualified them for primary endpoint analysis of sensitivity. MelaFind correctly identified 112/114 melanomas
Statistical Analysis 2: Comparison: Biopsied Pigmented Skin Lesions; Specificty of MelaFind and examining dermatologists on the same set of pigmented skin lesions; Test type: Superiority or Other; p = 0.02, Chi-squared

2. Secondary Outcome: Biopsy Ratio
Description: Number of lesions bioopsied to melanomas detected
Time Frame: Within 120 days of Data Lock
Reporting Status: Not Posted, anticipated posting 2009-12
Measure: Number

3. Secondary Outcome: Exploratory Analyses
Time Frame: Within 365 days of Data Lock
Reporting Status: Not Posted, anticipated posting 2010-02

ADVERSE EVENTS:
Arm/Group | Biopsied Pigmented Skin Lesions
Serious Adverse Events (participants affected / at risk) | 0/1383
Other Adverse Events (participants affected / at risk) | 0/1383

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days